CLINICAL TRIAL: NCT03003494
Title: Effectiveness and Handling of Spiolto® Respimat ® in COPD Patients - Italy
Acronym: OTIVACTO
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.43
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Spiolto® Respimat®: consented COPD patients who will be treated with Spiolto® Respimat® according to the approved SmPC
  Interventions: Drug: Spiolto® Respimat®

INTERVENTIONS:
Drug: Spiolto® Respimat® — observations taken in a period of approximately 6 weeks
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO

SUMMARY:
The purpose of the study is to measure changes in physical functioning in chronic obstructive pulmonary disease (COPD) patients being treated with Spiolto® Respimat® after approximately 6 weeks in routine clinical practice.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent prior to participation
2. Female and male patients = 40 years of age
3. Patients diagnosed with COPD and requiring long-acting dual bronchodilation (LAMA + LABA) treatment according to approved Spiolto® Respimat® SmPC and therapeutic plan recommendation

Exclusion criteria:

1. Patients with contraindications according to Spiolto® Respimat® Summary of Product Characteristics (SmPC)
2. Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 months
3. Patients continuing LABA-Inhalative Corticosteroids (ICS) treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists
4. Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
5. Pregnancy and lactation
6. Patients currently listed for lung transplantation
7. Current participation in any clinical trial or any other non-interventional study of a drug or device

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 chronic obstructive pulmonary disease (COPD) patients will be enrolled in Pulmonology sites
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (28):
- Italy (28):
  - Ospedale Generale Regionale "Miulli", Acquaviva Delle Fonti (BA)
  - Azienda Ospedaliera G. Rummo, Benevento
  - Casa di cura Mons. Calaciura, Biancavilla
  - Ospedale Orlandi, Bussolengo (VR)
  - IRCCS - Istituto Scientifico di Cassano delle Murge, Cassano Murge Bari
  - Università degli Studi "Magna Grecia" - Campus "S. Venuta", Catanzaro
  - Ospedale Mellino Mellini, Chiari (BS)
  - Osp. Piero Palagi, Florence
  - Ospedale Colonnello D Avanzo, Foggia
  - A.O. Ospedale Guido Salvini, Garbagnate Milanese
  - Presidio Ospedaliero di Imperia - ASL 1 Imperiese, Imperia
  - Ospedale della Versilia, LIDO DI Camaiore (LU)
  - Ospedale S. Salvatore, L’Aquila
  - Osp.dell'Angelo, Mestre
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Osp. dei Colli Monaldi-Cotugno, Napoli
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Ospedale S.Maria della Misericordia, AO di Perugia, Perugia
  - Azienda Ospedali Riuniti Marche Nord, Pesaro
  - Az.per Assist. Sanitaria N.5 Friuli Occidentale, Pordenone
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Università di Salerno, Salerno
  - Presidio Ospedaliero di Sesto S. Giovanni ASST Nord Milano, Sesto San Giovanni (MI)
  - Fondazione Salvatore Maugeri, Tradate (VA)
  - Ospedale di Cattinara, Trieste
  - Auxilium Vitae, Volterra

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carone M, Pennisi A, D'Amato M, Donati AF, Ricci A, Scognamillo C, Chun L, Aliani M, Ronsivalle V, Pelaia G. Physical Functioning in Patients with Chronic Obstructive Pulmonary Disease Treated with Tiotropium/Olodaterol Respimat in Routine Clinical Practice in Italy. Pulm Ther. 2020 Dec;6(2):261-274. doi: 10.1007/s41030-020-00122-9. Epub 2020 Jun 18. PMID 32557394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient with chronic Obstructive Pulmonary Disease receiving treatment Spiolto® Respimat® were enrolled between July 2017 and May 2018.
  309 screened and 3 patient violated inclusion/exclusion criteria were excluded, 306 entered the trial
Pre-assignment Details: All participants were screened for eligibility to participate in the study. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered if any one of the specific entry criteria were not met. Physical Functioning patient questionnaire (PF10)
Groups:
- Spiolto Respimat: Chronic Obstructive Pulmonary Disease (COPD) patients were administered a combination of tiotropium, an anticholinergic and olodaterol, a long-acting beta2-adrenergic agonist (LABA) in a Fixed dose combination through Respimat device according to approved Summary of Product Characteristics (SPC) and the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines
Period: Overall Study
Arm/Group | Spiolto Respimat
Started | 306
Completed | 278
Not Completed | 28
Not completed — Evaluable PF10 questionnaire at visit1 | 28

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The Treated set comprising all patients with informed consent, registration date and at least one documented administration of Spiolto® Respimat®.
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.04 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 216
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Therapeutic Success at Week 6 Approximately (Approx.) (Visit 2)
Description: Therapeutic success defined as at least 10-point increase of Physical functioning questionnaire (PF-10 ) score after approximately 6 weeks of Spiolto® Respimat® treatment The PF-10 used for assessing the primary outcome "physical functioning" is a sub-domain of the validated Short Form 36 (SF-36 ) and consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little" or "no, not limited at all", with a score of 1, 2 or 3. The sum of the scores of the 10 questions results in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "no, not limited at all"). The final sum of the individual scores was standardized to a range of 0 to 100 using the following formula: [(sum of scale items - 10) * 100] / 20. Higher scores indicate better physical functioning.
Time Frame: after approximately 6 weeks
Population: Full Analysis Set (FAS): The FAS comprised all patients of the Treated Set (TS) with a completed PF-10 questionnaire at both study visits.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 278
Percentage of Participants (%) | 52.52 [46.47 to 58.51]

2. Secondary Outcome: The Median Change in the PF-10 Score From Visit 1 (Baseline) to Visit 2
Description: The change in PF-10 score was determined by taking into account the individual change of each patient between Baseline (Visit 1) and Week 6 (approx.) (Visit 2) and then the median for change from baseline values across all subjects was calculated.
Time Frame: Baseline (visit 1) and after approx. week 6 (visit 2)
Population: FAS
Measure: Median (Full Range); unit: Unit on scale
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 278
Unit on scale | 10 [-60 to 80]

3. Secondary Outcome: Patients General Condition Evaluated by the Physician (PGE Score) at Visit 1 and Visit 2
Description: The patient's general condition was evaluated by means of Physician's Global Evaluation (PGE) score. The PGE score is documented on a scale from 1 (poor) to 8 (excellent) at both visits. 1-2: poor; 3-4: satisfactory; 5-6: good; 7-8: excellent
Time Frame: Baseline (visit 1) and after approx.week 6 (visit 2)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 278
Participants
  Baseline (Visit 1) : PGE score 1 | 2
  Baseline (Visit 1) : PGE score 2 | 5
  Baseline (Visit 1) : PGE score 3 | 69
  Baseline (Visit 1) : PGE score 4 | 72
  Baseline (Visit 1) : PGE score 5 | 65
  Baseline (Visit 1) : PGE score 6 | 46
  Baseline (Visit 1) : PGE score 7 | 19
  Baseline (Visit 1) : PGE score 8 | 0
  Week 6 (approx.) (Visit 2): Score 1 | 0
  Week 6 (approx.) (Visit 2): Score 2 | 2
  Week 6 (approx.) (Visit 2): Score 3 | 18
  Week 6 (approx.) (Visit 2): Score 4 | 32
  Week 6 (approx.) (Visit 2): Score 5 | 65
  Week 6 (approx.) (Visit 2): Score 6 | 113
  Week 6 (approx.) (Visit 2): Score 7 | 42
  Week 6 (approx.) (Visit 2): Score 8 | 6

4. Secondary Outcome: Patient Overall Satisfaction With Spiolto® Respimat®
Description: Patients were asked how overall satisfied they were with the Spiolto® Respimat® treatment at Week 6 (approx.) (Visit 2).
Time Frame: After approx. 6 weeks of treatment initiation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 278
Participants
  Very satisfied | 31
  Satisfied | 111
  Rather satisfied | 98
  Neither satisfied nor dissatisfied | 29
  Rather dissatisfied | 5
  Dissatisfied | 0
  Very dissatisfied | 2
  Questionnaire not completed | 2

5. Secondary Outcome: Patient Satisfaction With Inhaling From the Respimat® Device
Description: Patients were asked how satisfied they were by inhaling with the Respimat® device at Week 6 (approx.) (Visit 2)
Time Frame: After approx. 6 weeks of treatment initiation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 278
Participants
  Very satisfied | 47
  Satisfied | 119
  Rather satisfied | 83
  Neither satisfied nor dissatisfied | 23
  Rather dissatisfied | 2
  Dissatisfied | 1
  Very dissatisfied | 1
  Questionnaire not completed | 2

6. Secondary Outcome: Patient Satisfaction With Handling of the Respimat® Inhalation Device
Description: Patients were asked how satisfied they were with handling of the Respimat® inhalation device at Week 6 (approx.) (Visit 2).
Time Frame: After approx. 6 weeks of treatment initiation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto Respimat
Number analyzed (Participants) | 278
Participants
  Very satisfied | 57
  Satisfied | 121
  Rather satisfied | 70
  Neither satisfied nor dissatisfied | 19
  Rather dissatisfied | 4
  Dissatisfied | 5
  Very dissatisfied | 0
  Questionnaire not completed | 2

ADVERSE EVENTS:
Time Frame: From first drug administration until end of study, up to approx 6 weeks.
Description: All safety analyses were based on the TS
Arm/Group | Spiolto Respimat
All-Cause Mortality (participants affected / at risk) | 1/306
Serious Adverse Events (participants affected / at risk) | 2/306
Other Adverse Events (participants affected / at risk) | 0/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto Respimat (N=306)
Death (General disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Therapeutic success was assessed by a patient questionnaire at two time points. The respective answers were dependent on the condition of the patient at the completion. No objective assessment was performed due to the non-interventional study concept

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT03003494/SAP_000.pdf
  • Study Protocol (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03003494/Prot_001.pdf